CLINICAL TRIAL: NCT02631876
Title: FORWARD I: A Randomized, Open Label Phase 3 Study to Evaluate the Safety and Efficacy of Mirvetuximab Soravtansine (IMGN853) Versus Investigator's Choice of Chemotherapy in Women With Folate Receptor Alpha Positive Advanced Epithelial Ovarian Cancer, Primary Peritoneal Cancer or Fallopian Tube Cancer
Brief Title: A Study of Mirvetuximab Soravtansine vs. Investigator's Choice of Chemotherapy in Women With Folate Receptor (FR) Alpha Positive Advanced Epithelial Ovarian Cancer (EOC), Primary Peritoneal or Fallopian Tube Cancer
Acronym: FORWARD I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0403
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Ovarian Cancer
Keywords: Epithelial ovarian cancer; Fallopian tube cancer; Primary peritoneal cancer; IMGN853; ADC; Antibody drug conjugate; ImmunoGen; Antibody; Folate receptor alpha; mirvetuximab soravtansine; Phase 3; platinum-resistant; MIRV
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — mirvetuximab soravtansine; Paclitaxel; liposomal doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirvetuximab Soravtansine (Experimental): Participants will receive mirvetuximab soravtansine at 6 milligrams/kilogram (mg/kg) adjusted ideal body weight (AIBW) administered intravenously (IV) on Day 1 of a 3 week cycle. Participants will continue to receive study drug until they experience progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (as assessed by the blinded independent review committee [BIRC]), experience unacceptable toxicity, or withdraw consent, whichever comes first, or until the sponsor terminate the study. (Maximum exposure: 86.9 weeks)
  Interventions: Drug: Mirvetuximab soravtansine
- Investigator's Choice (IC) Chemotherapy (Experimental): Participants will receive a dose of IC chemotherapeutic agent calculated using body surface area (BSA). Paclitaxel will be administered at 80 milligrams/square meter (mg/m^2) as a 1-hour IV infusion on Days 1, 8, 15, and 22 of a 4-week cycle; or topotecan will be administered at 4 mg/m^2 over 30 minutes on Days 1, 8, and 15 of a 4-week cycle. Alternatively, topotecan could be administered at 1.25 mg/m^2 over 30 minutes on Days 1 to 5 of a 3-week cycle; or pegylated liposomal doxorubicin will be administered at 40 mg/m^2 as a 1 mg/minute IV infusion on Day 1 of a 4-week cycle. After Cycle 1, if tolerated, pegylated liposomal doxorubicin could be administered as a 1-hour infusion. Participants will continue to receive study drug until they experience PD per RECIST version 1.1 (as assessed by BIRC), experience unacceptable toxicity, or withdraw consent, whichever comes first, or until the sponsor terminate the study. (Maximum exposure: 62.9 weeks)
  Interventions: Drug: Paclitaxel; Drug: Pegylated liposomal doxorubicin; Drug: Topotecan

INTERVENTIONS:
Drug: Mirvetuximab soravtansine — Mirvetuximab Soravtansine will be administered per dose and schedule specified in the arm.
  Arms: Mirvetuximab Soravtansine
Drug: Paclitaxel — Paclitaxel will be administered per dose and schedule specified in the arm.
  Arms: Investigator's Choice (IC) Chemotherapy
Drug: Pegylated liposomal doxorubicin — Pegylated liposomal doxorubicin will be administered per dose and schedule specified in the arm.
  Arms: Investigator's Choice (IC) Chemotherapy
Drug: Topotecan — Topotecan will be administered per dose and schedule specified in the arm.
  Arms: Investigator's Choice (IC) Chemotherapy

SUMMARY:
This is a Phase 3, open label, randomized study designed to compare the safety and efficacy of mirvetuximab soravtansine to that of selected single-agent chemotherapy (Investigator's choice) in women with platinum-resistant FR-alpha positive advanced EOC, primary peritoneal cancer and/or fallopian tube cancer.

DETAILED DESCRIPTION:
Participants will be randomized to either mirvetuximab soravtansine or investigator's choice chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with advanced epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer
* Participants must have folate receptor alpha positive tumor expression as defined in the protocol
* Participants must have platinum-resistant ovarian cancer, defined as progression within 6 months from completion of a minimum of four cycles of platinum-containing therapy.
* Participants must have received at least one but no more than three prior systemic treatment regimens and for whom single-agent chemotherapy is appropriate as the next line of treatment
* Participants must have at least one lesion that meets the definition of measurable disease by RECIST 1.1

Exclusion Criteria:

* Diagnosis of clear cell, low grade ovarian cancer or mixed tumors
* Participants with primary platinum-refractory disease
* Serious concurrent illness or clinically relevant active infection as defined in the protocol
* Prior treatment with mirvetuximab soravtansine
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CMO ImmunoGen, Study Director — ImmunoGen, Inc.
Locations (131):
- United States (53):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - UCLA Women's Health Clinical Research Unit - OBGYN, Los Angeles, California
  - University of California San Diego Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Norwalk Hospital/WCHN, Norwalk, Connecticut
  - Florida State University College of Medicine, Sarasota, Florida
  - Georgia Regents University (GRU)-Medical College of Georgia (MCG) - Cancer Center, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Sudarshan Sharma LTD, Hinsdale, Illinois
  - Community Health Network, Inc., Indianapolis, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Women's Cancer Care, Covington, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - WK Physician Network Clinical Research, Shreveport, Louisiana
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mercy Women's Oncology, Springfield, Missouri
  - Center of Hope, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - MD Anderson Cancer Center - Cooper Health, Camden, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - The University of New Mexico Comprehensive Cancer Center - Memorial Medical Center, Albuquerque, New Mexico
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center and (MSK Monmouth) and ( MSK Westchester), New York, New York
  - Levine Cancer Institute - Carolinas Medical Center, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Fairview Hospital, Moll Pavilion Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Hillcrest Hospital, Mayfield, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee - Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Women & Infants of Rhode Island, Providence, Rhode Island
  - Hollings Cancer Center, Charleston, South Carolina
  - Texas Oncology-Austin Central, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Texas Oncology - The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Kadlec Clinic Hematology & Oncology, Kennewick, Washington
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Groeninge - Oncology Centre, Kortrijk
  - Universitaire Ziekenhuizen (UZ) Leuven-Gasthuisberg, Leuven
  - Centre Hospitalier de l'Ardenne, Libramont
- University Clinical Center of Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute - Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital de la CitedelaSante, Laval, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- Czechia (3):
  - Porodnicka A Gynekologicka Klinika, Hradec Králové
  - University Hospital Ostrava, Ostrava Poruba
  - Onkologicke oddeleni Krajske nemocnice T. Bati, a.s., Zlin, Zlín
- France (12):
  - Institut de Cancerologie de L'Ouest - site Paul Papin, Angers
  - CHRU Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Cochin Hospital, Paris
  - Hôpital Croix St-Simon, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Armoricain de radiotherapie, Imagerie Medicale et Oncol, Plérin
  - Centre Eugene Marquis, Rennes
  - Institut Curie-Hopital Rene Huguenin, Saint-Cloud
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy Institution, Villejuif
- Ireland (2):
  - Bon Secours Hospital, Cork
  - Mater Private Hospital and Mater Misericordiae University Hospital, Dublin
- Italy (9):
  - Istituto Europeo di Oncologia, Milan, MI
  - Azienda Ospedaliero Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Sanitaria Locale (ASL), Brindisi
  - Azienda Unita Sanitaria Locale di Ravenna, Faenza
  - Romagnolo per lo Studio e la Cura dei Tumori IRST-IRCCS - Oncologia medica, Meldola (FC)
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS National Cancer Institute, Milan
  - Istituto Nazionale Tumori- G. Pascale, Naples
  - Policlinico Universitario Agostino Gemelli, Roma
- Russia (4):
  - LLC "VitaMed", Moscow
  - State Budget-Funded Healthcare Institution of Novosibirsk Oblast "Novosibirsk Oblast Oncology Dispensary", Novosibirsk
  - Budget-Funded Healthcare Institution of Omsk Oblast "Clinical Oncology Dispensary", Omsk
  - State Budget Institution of Health "Leningrad Regional Oncologicacal Dispensary", Saint Petersburg
- Serbia (3):
  - Oncology and Radiology Institute Serbia, Belgrade
  - Oncology Institute Vojvodina, Kamenitz
  - Clinical Centre Nis, Oncology Clinic, Niš
- Spain (16):
  - ICO Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Gipuzkoa
  - Hospital Teresa Herrera (CHUACoruña), A Coruña
  - IOR - Hospital Quiron Dexeus, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Institut Català d'Oncologia - Unitad de Investigación Clínica, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Complejo Hospitalario Granada, Granada
  - Hospital Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center - Madrid, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Servicio de Oncología Médica Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario Malaga - Hospital Materno Infantil de Málaga, Málaga
  - Hospital Son Llatzer (HSLL), Palma de Mallorca
  - Instituto Valenciano de Oncologia, Valencia
- Switzerland (3):
  - Kantonsspital Winterthur, Medizinische Onkologie, Winterthur, Canton of Zurich
  - Kantonsspital, Winterthur, Canton of Zurich
  - Hopitaux Universitaires de Geneve, Geneva
- United Kingdom (11):
  - UCL Cancer Institute, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham, England
  - Lancashire Teaching Hospitals NHS Foundation Trust - Royal Preston Hospital, Preston, England
  - The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital (RMH), Sutton, England
  - The Royal Wolverhampton Hospitals NHS Trust - New Cross Hospital - GOW, Wolverhampton, England
  - Peterborough City Hospital, Peterborough, Great Britain
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Cancer,Haematology and Physics Directorate, Cancer Centre Royal Stoke University, Stoke-on-Trent, Staffordshire
  - University Hospitals Coventry & Warwickshire NHS Trust, Arden Cancer Centre, Coventry
  - Mount Vernon Cancer Centre, Northwood

REFERENCES:
- [Derived] Moore KN, Oza AM, Colombo N, Oaknin A, Scambia G, Lorusso D, Konecny GE, Banerjee S, Murphy CG, Tanyi JL, Hirte H, Konner JA, Lim PC, Prasad-Hayes M, Monk BJ, Pautier P, Wang J, Berkenblit A, Vergote I, Birrer MJ. Phase III, randomized trial of mirvetuximab soravtansine versus chemotherapy in patients with platinum-resistant ovarian cancer: primary analysis of FORWARD I. Ann Oncol. 2021 Jun;32(6):757-765. doi: 10.1016/j.annonc.2021.02.017. Epub 2021 Mar 2. PMID 33667670

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 366 participants were randomized in 2:1 to receive either mirvetuximab soravtansine or the investigator's choice (IC) chemotherapy.
Groups:
- Mirvetuximab Soravtansine: Participants received mirvetuximab soravtansine at 6 milligrams/kilogram (mg/kg) adjusted ideal body weight (AIBW) administered intravenously (IV) on Day 1 of a 3 week cycle. Participants continued to receive study drug until they experienced progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (as assessed by the blinded independent review committee [BIRC]), experienced unacceptable toxicity, or withdrew consent, whichever came first, or until the sponsor terminated the study. (Maximum exposure: 86.9 weeks)
- Investigator's Choice (IC) Chemotherapy: Participants received a dose of IC chemotherapeutic agent calculated using body surface area (BSA). Paclitaxel administered at 80 milligrams/square meter (mg/m^2) as a 1-hour IV infusion on Days 1, 8, 15, and 22 of a 4-week cycle; or topotecan administered at 4 mg/m^2 over 30 minutes on Days 1, 8, and 15 of a 4-week cycle. Alternatively, topotecan could have been administered at 1.25 mg/m^2 over 30 minutes on Days 1 to 5 of a 3-week cycle; or pegylated liposomal doxorubicin administered at 40 mg/m^2 as a 1 mg/minute IV infusion on Day 1 of a 4-week cycle. After Cycle 1, if tolerated, pegylated liposomal doxorubicin could have been administered as a 1-hour infusion. Participants continued to receive study drug until they experienced PD per RECIST version 1.1 (as assessed by BIRC), experienced unacceptable toxicity, or withdrew consent, whichever came first, or until the sponsor terminated the study. (Maximum exposure: 62.9 weeks)
Period: Overall Study
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Started (ITT population: all participants randomized in the study.) | 248 | 118
Safety Population (Enrolled participants who received at least 1 dose of mirvetuximab soravtansine or IC chemotherapy.) | 243 | 109
Completed | 129 | 55
Not Completed | 119 | 63
Not completed — Death | 96 | 50
Not completed — Investigator's discretion | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Other than specified | 4 | 4

BASELINE CHARACTERISTICS:
Population: ITT population included all participants randomized in the study.
Groups:
- Mirvetuximab Soravtansine: Participants received mirvetuximab soravtansine at 6 mg/kg AIBW administered IV on Day 1 of a 3 week cycle. Participants continued to receive study drug until they experienced PD per RECIST version 1.1 (as assessed by BIRC), experienced unacceptable toxicity, or withdrew consent, whichever came first, or until the sponsor terminated the study. (Maximum exposure: 86.9 weeks)
- Investigator's Choice (IC) Chemotherapy: Participants received a dose of IC chemotherapeutic agent calculated using BSA. Paclitaxel administered at 80 mg/m^2 as a 1-hour IV infusion on Days 1, 8, 15, and 22 of a 4-week cycle; or topotecan administered at 4 mg/m^2 over 30 minutes on Days 1, 8, and 15 of a 4-week cycle. Alternatively, topotecan could have been administered at 1.25 mg/m^2 over 30 minutes on Days 1 to 5 of a 3-week cycle; or pegylated liposomal doxorubicin administered at 40 mg/m^2 as a 1 mg/minute IV infusion on Day 1 of a 4-week cycle. After Cycle 1, if tolerated, pegylated liposomal doxorubicin could have been administered as a 1-hour infusion. Participants continued to receive study drug until they experienced PD per RECIST version 1.1 (as assessed by BIRC), experienced unacceptable toxicity, or withdrew consent, whichever came first, or until the sponsor terminated the study. (Maximum exposure: 62.9 weeks)
- Total: Total of all reporting groups
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy | Total
Number analyzed (Participants) | 248 | 118 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.29) | 62.9 (10.51) | 62.8 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 118 | 366
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 225 | 102 | 327
  Unknown or Not Reported | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 225 | 105 | 330
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), as Assessed by BIRC Per RECIST Version 1.1 in All Participants Randomized to the Study
Description: PFS was defined as the time from randomization until PD or death whichever occurred first, estimated using the Kaplan-Meier method. PD: At least a 20% increase in the sum of the longest diameters (SoD) of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: From the date of randomization until the time of death or PD (maximum exposure: 86.9 weeks for mirvetuximab soravtansine arm and 62.9 weeks for IC chemotherapy arm)
Population: ITT population included all participants randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 248 | 118
months | 4.14 [3.75 to 4.53] | 4.44 [2.83 to 5.59]

2. Primary Outcome: PFS, as Assessed by BIRC Per RECIST Version 1.1 in Participants With High Folate Receptor Alpha Level (≥ 75% of Tumor Staining)
Description: PFS was defined as the time from randomization until PD or death whichever occurred first, estimated using the Kaplan-Meier method. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: as for outcome 1
Population: ITT population included all participants randomized in the study. Here, overall number of participants analyzed signifies participants with high folate receptor alpha level.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 147 | 71
months | 4.76 [4.11 to 5.68] | 3.25 [1.97 to 5.59]

3. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response, as Assessed by BIRC Per RECIST1.1
Description: ORR was defined as percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR: At least 30 percent (%) decrease in the SoD of target lesions, taking as reference the baseline SoD.
Time Frame: From randomization until first BOR of CR or PR (maximum exposure: 86.9 weeks for mirvetuximab soravtansine arm and 62.9 weeks for IC chemotherapy arm)
Population: ITT population included all participants randomized in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 248 | 118
percentage of participants | 22 [17.2 to 27.9] | 12 [6.6 to 19.1]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause. Participants who did not experience the event of death were censored at their last date known to be alive. OS was estimated using the Kaplan-Meier method.
Time Frame: From the date of randomization until the time of death (maximum exposure: 86.9 weeks for mirvetuximab soravtansine arm and 62.9 weeks for IC chemotherapy arm)
Population: ITT population included all participants randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 248 | 118
months | 15.57 [12.85 to 18.04] | 13.93 [11.40 to 18.50]

5. Secondary Outcome: Number of Participants Achieving at Least a 15% (≥ 15-Point) Absolute Improvement From Baseline on the EORTC QLQ-OV28 Abdominal/Gastrointestinal (AB/GI) Symptom Subscale at Week 8/9 Assessment
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Ovarian Cancer 28 (EORTC QLQ-OV28) is a 28-item ovarian cancer supplemental module. It comprises of 6 symptom scales (AB/GI symptoms, peripheral neuropathy, other chemotherapy side-effects, hormonal symptoms, body image, attitude to disease, treatment), and sexual functioning. Participants were asked to indicate extent to which they experienced AB/GI symptoms. Participants responded on a scale of 1-4(1=not at all, 2=a little, 3=quite a bit, 4=very much) to following: Did you have abdominal pain? Did you have a bloated feeling in your abdomen? Did you have problems with your clothes feeling too tight? Did you experience any change in bowel habit as a result of your disease or treatment? Were you troubled by passing wind/gas/flatulence? Have you felt full too quickly after beginning to eat? Have you had indigestion/heartburn? Data were transformed to a scale from 0-100. Lower scores=better health.
Time Frame: Baseline, Week 8/9
Population: ITT population included all participants randomized in the study. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 142 | 50
Participants | 45 | 7

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE): any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to study drug. Severity: graded per National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) v4.03 on following scale: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening, Grade 5=death. Relation of AE to treatment was determined by investigator. Serious AEs: death, life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent/significant disability or incapacity, congenital anomaly or birth defect, or an important medical event that required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs: any AE that emerged on or after the first dose, and within 30 days of the last dose. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported AEs module.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 86.9 weeks for mirvetuximab soravtansine arm and 62.9 weeks for IC chemotherapy arm)
Population: Safety population included all enrolled participants who received at least 1 dose of mirvetuximab soravtansine or IC chemotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 243 | 109
Participants | 242 | 107

7. Secondary Outcome: Gynecologic Cancer Intergroup (GCIG) CA-125 Response Rate: Percentage of Participants With GCIG CA-125 Confirmed Clinical Responses
Description: CA-125 Response rate wasdefined as the number of participants with a CA-125 confirmed response divided by the number of participants in the CA-125 response-evaluable population multiplied by 100.
Time Frame: From first dose of study drug until CA-125 response (maximum exposure: 86.9 weeks for mirvetuximab soravtansine arm and 62.9 weeks for IC chemotherapy arm)
Population: CA-125-Evaluable population included all randomized population whose pretreatment sample was ≥ 2.0 times the upper limit of normal (ULN), within 2 weeks prior to randomization, and who had at least 1 post-baseline CA 125 evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Mirvetuximab Soravtansine: Participants received MIRV mirvetuximab soravtansine at 6 mg/kg AIBW administered IV on Day 1 of a 3 week cycle. Participants continued to receive study drug until they experienced PD per RECIST version 1.1 (as assessed by BIRC), experienced unacceptable toxicity, or withdrew consent, whichever came first, or until the sponsor terminated the study. (Maximum exposure: 86.9 weeks)
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 203 | 82
percentage of participants | 51 [44.1 to 58.3] | 27 [17.6 to 37.8]

8. Secondary Outcome: PFS, as Assessed by Investigator Per RECIST Version 1.1
Description: as for outcome 2
Time Frame: as for outcome 1
Population: ITT population included all participants randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 248 | 118
months | 4.27 [4.11 to 5.06] | 4.24 [2.76 to 5.36]

9. Secondary Outcome: Duration of Response (DOR), as Assessed by BIRC Per RECIST v1.1
Description: DOR was defined as the time from the date of the first response (CR or PR), whichever was recorded first, until the date of PD. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase. DOR was only defined for participants who had a BOR of CR or PR using the method of Kaplan-Meier.
Time Frame: From the date of first response (CR or PR) until the date of PD (maximum exposure: 86.9 weeks for mirvetuximab soravtansine arm and 62.9 weeks for IC chemotherapy arm)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 55 | 14
months | 5.65 [4.17 to 8.51] | 7.26 [4.14 to NA] — Data not calculated due to less number of participants with an event

10. Secondary Outcome: Area Under the Plasma Concentration-Versus Time Curve From Time of Dose Until Tlast (AUClast) of Mirvetuximab Soravtansine,Total M9346A Antibody, DM4, and S-methyl DM4
Description: PK parameters were calculated using standard non-compartmental methods.
Time Frame: Pre-dose and within 5 minutes after mirvetuximab soravtansine infusion on Day 1 of Cycles 1 and 3; and Day 8 and 15 of Cycles 1 and 3
Population: PK population included all participants who received at least 1 infusion of mirvetuximab soravtansine, had evaluable PK data, and had samples collected with no major deviations related to administration of study drug. Here, 'number analyzed'=participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: hours*milligrams/milliliter (hr*mg/mL)
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 235
hours*milligrams/milliliter (hr*mg/mL)
  Mirvetuximab Soravtansine at Cycle 1 | 20.53 (10.31)
  Mirvetuximab Soravtansine at Cycle 3: number analyzed (Participants) | 146
  Mirvetuximab Soravtansine at Cycle 3 | 22.40 (7.770)
  Total M9346A antibody at Cycle 1 | 23.23 (9.463)
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 146
  Total M9346A antibody at Cycle 3 | 31.20 (11.52)
  DM4 at Cycle 1: number analyzed (Participants) | 233
  DM4 at Cycle 1 | 348.5 (265.7)
  DM4 at Cycle 3: number analyzed (Participants) | 142
  DM4 at Cycle 3 | 347.4 (280.9)
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 234
  S-methyl DM4 at Cycle 1 | 1586 (1496)
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 146
  S-methyl DM4 at Cycle 3 | 1512 (1278)

11. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA)
Description: An electrochemiluminescent method was used for the detection of anti-mirvetuximab soravtansine antibodies in plasma from samples collected in dipotassium ethylenediaminetetraacetic acid (K2EDTA) tubes. The qualitative assay was designed to detect anti-mirvetuximab soravtansine antibodies in human plasma.
Time Frame: Pre-dose and within 5 minutes after mirvetuximab soravtansine infusion on Day 1 of Cycles 1, 2, and 4; pre-dose on Day 1 of Cycle 6
Population: Immunogenicity population included all participants who received at least 1 infusion of mirvetuximab soravtansine and had evaluable immunogenicity data.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvetuximab Soravtansine
Number analyzed (Participants) | 230
Participants | 13

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 86.9 weeks for mirvetuximab soravtansine arm and 62.9 weeks for IC chemotherapy arm)
Description: Safety population included all enrolled participants who received at least 1 dose of mirvetuximab soravtansine or IC chemotherapy.
Arm/Group | Mirvetuximab Soravtansine | Investigator's Choice (IC) Chemotherapy
All-Cause Mortality (participants affected / at risk) | 96/243 | 50/109
Serious Adverse Events (participants affected / at risk) | 67/243 | 31/109
Other Adverse Events (participants affected / at risk) | 242/243 | 106/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvetuximab Soravtansine (N=243) | Investigator's Choice (IC) Chemotherapy (N=109)
Intestinal obstruction (Gastrointestinal disorders) | 10 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 4 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 2 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Oesophageal infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Systemic infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Complication associated with device (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Eye pain (Eye disorders) | 1 | 0
Punctate keratitis (Eye disorders) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvetuximab Soravtansine (N=243) | Investigator's Choice (IC) Chemotherapy (N=109)
Nausea (Gastrointestinal disorders) | 131 | 46
Diarrhoea (Gastrointestinal disorders) | 107 | 18
Abdominal pain (Gastrointestinal disorders) | 80 | 23
Constipation (Gastrointestinal disorders) | 64 | 31
Vomiting (Gastrointestinal disorders) | 64 | 22
Abdominal distension (Gastrointestinal disorders) | 26 | 11
Dyspepsia (Gastrointestinal disorders) | 18 | 5
Abdominal pain upper (Gastrointestinal disorders) | 15 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 5
Dry mouth (Gastrointestinal disorders) | 11 | 2
Abdominal pain lower (Gastrointestinal disorders) | 10 | 3
Stomatitis (Gastrointestinal disorders) | 10 | 23
Ascites (Gastrointestinal disorders) | 9 | 6
Abdominal discomfort (Gastrointestinal disorders) | 8 | 0
Flatulence (Gastrointestinal disorders) | 7 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Aphthous ulcer (Gastrointestinal disorders) | 3 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 1
Retching (Gastrointestinal disorders) | 3 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1
Abnormal faeces (Gastrointestinal disorders) | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0
Coating in mouth (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Faecal vomiting (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Rectal discharge (Gastrointestinal disorders) | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0
Vomiting projectile (Gastrointestinal disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 2
Glossitis (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Tongue pigmentation (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 83 | 38
Asthenia (General disorders) | 51 | 25
Pyrexia (General disorders) | 25 | 7
Non-cardiac chest pain (General disorders) | 9 | 1
Oedema peripheral (General disorders) | 8 | 10
Chills (General disorders) | 7 | 2
Peripheral swelling (General disorders) | 6 | 1
Influenza like illness (General disorders) | 4 | 6
Malaise (General disorders) | 4 | 1
Pain (General disorders) | 4 | 3
Chest discomfort (General disorders) | 3 | 0
Adverse drug reaction (General disorders) | 2 | 0
Chest pain (General disorders) | 2 | 1
Cyst (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 2
Injection site bruising (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 2 | 6
Catheter site erythema (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Early satiety (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Hernia pain (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0
Infusion site reaction (General disorders) | 1 | 0
Injection site swelling (General disorders) | 1 | 0
Catheter site inflammation (General disorders) | 0 | 1
Catheter site rash (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Vision blurred (Eye disorders) | 104 | 6
Keratopathy (Eye disorders) | 77 | 1
Dry eye (Eye disorders) | 68 | 2
Visual acuity reduced (Eye disorders) | 52 | 2
Cataract (Eye disorders) | 36 | 2
Photophobia (Eye disorders) | 34 | 2
Eye pain (Eye disorders) | 31 | 1
Vitreous floaters (Eye disorders) | 13 | 0
Foreign body sensation in eyes (Eye disorders) | 9 | 0
Visual impairment (Eye disorders) | 9 | 1
Keratitis (Eye disorders) | 8 | 0
Eye irritation (Eye disorders) | 7 | 0
Lacrimation increased (Eye disorders) | 6 | 1
Corneal deposits (Eye disorders) | 5 | 0
Eye pruritus (Eye disorders) | 5 | 0
Ocular discomfort (Eye disorders) | 5 | 1
Punctate keratitis (Eye disorders) | 4 | 0
Blepharitis (Eye disorders) | 3 | 0
Diplopia (Eye disorders) | 3 | 0
Glaucoma (Eye disorders) | 3 | 0
Photopsia (Eye disorders) | 3 | 0
Uveitis (Eye disorders) | 3 | 0
Asthenopia (Eye disorders) | 2 | 0
Chalazion (Eye disorders) | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Conjunctival hyperaemia (Eye disorders) | 2 | 0
Lacrimation decreased (Eye disorders) | 2 | 0
Metamorphopsia (Eye disorders) | 2 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0
Xerophthalmia (Eye disorders) | 2 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0
Acquired corneal dystrophy (Eye disorders) | 1 | 0
Age-related macular degeneration (Eye disorders) | 1 | 0
Blepharochalasis (Eye disorders) | 1 | 0
Cataract nuclear (Eye disorders) | 1 | 0
Conjunctival irritation (Eye disorders) | 1 | 0
Corneal cyst (Eye disorders) | 1 | 0
Corneal oedema (Eye disorders) | 1 | 0
Dyschromatopsia (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Eye inflammation (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Eyelid pain (Eye disorders) | 1 | 0
Eyelid skin dryness (Eye disorders) | 1 | 0
Halo vision (Eye disorders) | 1 | 0
Hypermetropia (Eye disorders) | 1 | 0
Meibomianitis (Eye disorders) | 1 | 0
Myopia (Eye disorders) | 1 | 0
Night blindness (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Ocular toxicity (Eye disorders) | 1 | 0
Optic nerve disorder (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 1 | 0
Pupils unequal (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinal drusen (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Sympathetic ophthalmia (Eye disorders) | 1 | 0
Trichiasis (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Headache (Nervous system disorders) | 57 | 14
Neuropathy peripheral (Nervous system disorders) | 48 | 8
Dysgeusia (Nervous system disorders) | 30 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 11
Dizziness (Nervous system disorders) | 16 | 3
Paraesthesia (Nervous system disorders) | 15 | 5
Neurotoxicity (Nervous system disorders) | 9 | 6
Hypoaesthesia (Nervous system disorders) | 5 | 0
Sciatica (Nervous system disorders) | 4 | 0
Syncope (Nervous system disorders) | 3 | 0
Balance disorder (Nervous system disorders) | 2 | 0
Disturbance in attention (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 2 | 0
Neuralgia (Nervous system disorders) | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 1
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 0
Sensorimotor disorder (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Ageusia (Nervous system disorders) | 0 | 1
Drooling (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 60 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 40 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 4
Dehydration (Metabolism and nutrition disorders) | 9 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | 16
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 43 | 8
Alanine aminotransferase increased (Investigations) | 40 | 6
Blood alkaline phosphatase increased (Investigations) | 19 | 4
Weight decreased (Investigations) | 17 | 4
Gamma-glutamyltransferase increased (Investigations) | 7 | 1
Blood creatinine increased (Investigations) | 6 | 2
Transaminases increased (Investigations) | 5 | 0
Intraocular pressure increased (Investigations) | 4 | 0
Weight increased (Investigations) | 4 | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Urine leukocyte esterase positive (Investigations) | 2 | 0
Alanine aminotransferase (Investigations) | 1 | 0
Blood alkaline phosphatase (Investigations) | 1 | 0
Blood chloride decreased (Investigations) | 1 | 1
Blood creatine increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine (Investigations) | 1 | 0
Blood fibrinogen increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood iron decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0
Intestinal transit time decreased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Mean cell haemoglobin decreased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Urobilinogen urine increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1
Carbohydrate antigen 125 increased (Investigations) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
Procalcitonin increased (Investigations) | 0 | 1
Urinary tract infection (Infections and infestations) | 28 | 11
Nasopharyngitis (Infections and infestations) | 11 | 4
Upper respiratory tract infection (Infections and infestations) | 9 | 3
Cystitis (Infections and infestations) | 7 | 3
Influenza (Infections and infestations) | 6 | 3
Conjunctivitis (Infections and infestations) | 5 | 5
Respiratory tract infection (Infections and infestations) | 5 | 3
Pharyngitis (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 1
Ear infection (Infections and infestations) | 2 | 0
Gingivitis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Candida infection (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Keratitis bacterial (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 1
Oral fungal infection (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyuria (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Application site folliculitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 2
Nasal herpes (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 34 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 17
Neutropenia (Blood and lymphatic system disorders) | 16 | 43
Leukopenia (Blood and lymphatic system disorders) | 9 | 16
Lymphopenia (Blood and lymphatic system disorders) | 8 | 3
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Granulomatous lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 7
Rash (Skin and subcutaneous tissue disorders) | 10 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 14
Erythema (Skin and subcutaneous tissue disorders) | 7 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 4
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 16
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 5
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 2
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 4
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 4
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 23 | 16
Anxiety (Psychiatric disorders) | 14 | 8
Depression (Psychiatric disorders) | 6 | 2
Agitation (Psychiatric disorders) | 2 | 1
Depressed mood (Psychiatric disorders) | 2 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Tangentiality (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 16 | 4
Flushing (Vascular disorders) | 8 | 1
Hot flush (Vascular disorders) | 6 | 3
Haematoma (Vascular disorders) | 3 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 2
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 2
Varicose vein (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 7 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 4
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 1
Abdominal wall wound (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Haematuria (Renal and urinary disorders) | 7 | 2
Pollakiuria (Renal and urinary disorders) | 6 | 1
Dysuria (Renal and urinary disorders) | 5 | 4
Micturition urgency (Renal and urinary disorders) | 4 | 0
Urinary incontinence (Renal and urinary disorders) | 4 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bladder irritation (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 1
Dyspareunia (Reproductive system and breast disorders) | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Vulva cyst (Reproductive system and breast disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 8 | 2
Palpitations (Cardiac disorders) | 3 | 2
Sinus tachycardia (Cardiac disorders) | 3 | 2
Arrhythmia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 2
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Infusion related reaction (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Wound drainage (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT02631876/SAP_000.pdf
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02631876/Prot_001.pdf